CLINICAL TRIAL: NCT03181880
Title: To Evaluate Effectiveness of Aclidinium Bromide/Formoterol Fumarate Dihydrate in Chronic Obstructive Pulmonary Disease
Acronym: ASTUTE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped early as AZ have re-prioritised to focus on research to help bring existing and innovative medicines to more patients with asthma and COPD.
Sponsor: AstraZeneca (Industry)
Collaborators: QuintilesIMS, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6570R00004
Record Dates: First submitted 2017-04-26; First posted 2017-06-09 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: ASTUTE; Chronic Obstructive Pulmonary Disease; Randomised; Pragmatic; Standard of Care; Aclidinium bromide/formoterol fumarate fixed-dose combination; Duaklir; Genuair
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aclidinium/formoterol (Active Comparator): Patients will be randomized to receive either Aclidinium bromide/formoterol fumarate fixed-dose combination
  Interventions: Drug: Aclidinium bromide/formoterol fumarate combination
- Bronchodilators (Active Comparator): The comparator arm consists of SOC.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Aclidinium bromide/formoterol fumarate combination — Patients will be randomized to receive either Aclidinium bromide/formoterol fumarate fixed-dose combination (Duaklir™ Genuair®), or Standard Of Care (SOC) Bronchodilators.
  The product in study is Aclidinium bromide/formoterol fumarate fixed-dose combination (Duaklir™ Genuair®).
  Each inhaler will contain at least 60 doses (and a maximum of 68 doses) of aclidinium bromide/formoterol fixed-dose combination 400μg /12μg. Patients will be instructed to take 1 puff in the morning (09:00 ± 1 h) and 1 puff in the evening (21:00 ± 1 h) during the 12 weeks of treatment.
  Other Names: Duaklir™ Genuair®
  Arms: Aclidinium/formoterol
Drug: Standard of Care — Brochodilators
  Arms: Bronchodilators

SUMMARY:
ASTUTE is a pragmatic open randomised 12-week multinational trial to evaluate the effectiveness of aclidinium bromide/formoterol fumarate dihydrate fixed-dose combination compared to standard of care bronchodilators in chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
ASTUTE is a longitudinal, randomised, multicentre, and multinational pragmatic study of patients with Chronic Obstructive Pulmonary Disease to evaluate the comparative effectiveness of Aclidinium bromide/formoterol fumarate fixed-dose combination (Duaklir™ Genuair®) and Standard of Care bronchodilators in patients treated with long acting bronchodilator monotherapies OR patients who abide to the following treatment category: patient is newly diagnosed, or naïve to maintenance therapy, or treated with short-acting bronchodilators as rescue medication, or has not been treated with long-acting bronchodilators in the last 3 months.

ELIGIBILITY:
Inclusion Criteria:

Patient is aged 40 years or older;

* Confirmed diagnosis of COPD;
* Spirometry performed at study entry or within the last 3 months preceding study entry with a post-bronchodilator Forced Expiratory Volume in 1 Second/Forced Vital Capacity quotient less than 0.7;
* Patient is a current smoker or an ex-smoker with a smoking history of ≥10 pack-years;
* Patient belongs to any of these treatment groups:

  * Patient is treated by a monotherapy long-acting bronchodilator (Long-Acting Muscarinic Antagonist or Long-Acting Beta Agonist), or
  * Naïve COPD patient, defined as:
* Patient is newly diagnosed, or
* Patient is naïve to maintenance therapy, or
* Patient is treated with short acting bronchodilators as rescue medication, or
* Patient has not been treated with long acting bronchodilators in the last 3 months.

Exclusion Criteria:

-

Patients should not be included in the study if any of the following exclusion criteria applies:

* Patient changed COPD treatment regimen over the preceding 3 months;
* Patient treated or intended to be treated at the time of randomisation with a maintenance regimen of inhaled corticosteroids or inhaled corticosteroids-containing medications;
* Patient treated or intended to be treated at the time of randomisation with aclidinium bromide/formoterol fumarate dihydrate inhalation powder;
* Patient had a previous diagnosis of asthma or is suspected of having asthma, asthma-COPD overlap or any other chronic respiratory disease other than COPD (including severe ones, such as cystic fibrosis, pulmonary fibrosis, active neoplasm except adequately treated [no evidence of recurrence within 5 years], active tuberculosis);
* Patient developed a respiratory tract infection or COPD exacerbation within 6 weeks (or 3 months if an exacerbation-related hospitalisation was required) before the randomisation visit;
* Patient with a history of hypersensitivity reaction to inhaled anticholinergics, sympathomimetic amines, lactose monohydrate, inhaled medication, or any component thereof (including report of paradoxical bronchospasm);
* Patient has been previously enrolled in the current study.
* Any condition that in the Investigator's opinion, would limit a patient's ability to participate in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-04 (Estimated); Primary Completion 2018-12-03 (Estimated); Study Completion 2018-12-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in overall early morning COPD symptom severity score of aclidinium bromide/formoterol fumarate dihydrate inhalation powder vs. Standard of Care bronchodilators as measured by the Early Morning Symptoms of COPD Instrument over 12 wks. | study entry and previous day (retrospectively), days 22-28, days 50-56, days 78-84
  Changes from baseline compared between aclidinium bromide/formoterol fumarate dihydrate inhalation powder and Standard of Care bronchodilators. Baseline values for EMSCI will be averaged over the study entry and previous day. For longitudinal analyses, each daily measure will be aggregated on a weekly (7 days) basis during the weeks of measurement (weeks 4, 8, and/or 12) by taking the mean value of all available measurements during the week.
Change from baseline in overall night time COPD symptom severity score of aclidinium bromide/formoterol fumarate dihydrate inhalation powder vs. Standard of Care bronchodilators as measured by the Nighttime Symptoms of COPD Instrument over 12 weeks. | study entry and previous day (retrospectively), days 22-28, days 50-56, days 78-84
  Changes from baseline compared between aclidinium bromide/formoterol fumarate dihydrate inhalation powder and Standard of Care bronchodilators. Baseline values for NiSCI will be averaged over the study entry and previous day. For longitudinal analyses, each daily measure will be aggregated on a weekly (7 days) basis during the weeks of measurement (weeks 4, 8, and/or 12) by taking the mean value of all available measurements during the week.

SECONDARY OUTCOMES:
Change from baseline in daily RS total Score of aclidinium bromide/formoterol fumarate dihydrate inhalation powder versus Standard of Care bronchodilators measured by the E-RS™COPD scale over 12 weeks. | study entry and previous day (retrospectively), days 22-28, days 50-56, days 78-84
  Baseline values of the RS-Total Score will be collected and averaged at the study entry visit and previous day.
  The secondary effectiveness variable will be estimated by the change from baseline in daily RS-Total Score over 12 weeks of treatment.
Change from baseline in health status of aclidinium bromide/formoterol fumarate dihydrate inhalation powder versus Standard of Care bronchodilatorsmeasured by the COPD assessment Test (CAT) over 12 weeks. | study entry, days 28, 56 and 84
  The CAT measures the health status of patients with COPD. If the response to 1 of the 8 items is missing, the score will be considered missing. Change from baseline in health status over 12 weeks of follow-up (on the last day of weeks 4, 8, and 12) will be calculated. These change scores will be the CAT endpoint.
Change from baseline in total time index of aclidinium bromide/formoterol fumarate dihydrate inhalation powder versus Standard of Care bronchodilators measured by the Yale Physical Activity Survey (YPAS) over 12 weeks. | study entry, days 28, 56 and 84
  The Total Time Index will be calculated at baseline and over 12 weeks of follow-up (on the last day of weeks 4, 8, and 12). Change from baseline will be calculated. These change scores will be the Total Time Index analysed.
Change from baseline in Energy Expenditure Index of aclidinium bromide/formoterol fumarate dihydrate inhalation powder versus Standard of Care bronchodilators measured by the Yale Physical Activity Survey (YPAS) over 12 weeks. | study entry, days 28, 56 and 84
  The Energy Expenditure Index will be calculated at baseline and over 12 weeks of follow-up (on the last day of weeks 4, 8, and 12). Change from baseline will be calculated. These change scores will be the Energy Expenditure Index analysed.
Change from baseline in Activity Dimensions Summary Index of aclidinium bromide/formoterol fumarate dihydrate inhalation powder versus Standard of Care bronchodilators measured by the Yale Physical Activity Survey (YPAS) over 12 weeks. | study entry, days 28, 56 and 84
  The Activity Dimensions Summary Index will be calculated at baseline and over 12 weeks of follow-up (on the last day of weeks 4, 8, and 12). Change from baseline will be calculated. These change scores will be the Activity Dimensions Summary Index analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ribera, Study Director — AstraZeneca

IPD SHARING:
Plan to Share IPD: No